CLINICAL TRIAL: NCT06272422
Title: Comparison of the Restoration of Hip Biomechanical Parameters by CT Measurement Between the 3 Surgical Techniques: RSA/Minihip/THA
Brief Title: Comparison of the Restoration of Hip Biomechanical Parameters by CT Measurement Between the 3 Surgical Techniques: RSA/Minihip/THA - Hip Replacement: 3D Planning
Acronym: HIP3D
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/0472; 2023-A00358-37 (Other: IDRCB - ANSM ID)
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Coxarthrosis
Keywords: Arthroplasty hip; femoral offset; resurfacing; EOS; 3D
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- total hip arthroplasty (THA): Standard THA, the head and neck of the femur are cut.
  Interventions: Procedure: hip arthroplasty
- Total hip prosthesis with femoral neck preservation: A total hip replacement is performed, but the neck of the femur is preserved and the head of the femur is cut off.
  Interventions: Procedure: hip arthroplasty
- Hip resurfacing: the head and neck of the femur are preserved.
  Interventions: Procedure: hip arthroplasty

INTERVENTIONS:
Procedure: hip arthroplasty — resurfacing procedures (HRP), THA and Minihip-type neck-preserving total hip arthroplasty.

SUMMARY:
The study will analyze hip biomechanical parameters using EOS radiographic measurements pre- and post-operatively (3 months) and post-operatively (3 months) CT scans after total hip replacement (THR), neck-preserving THR of the Minihip type or hip resurfacing (HR). Clinical results will be assessed at 3 months and 1 year after surgery.

To this end, two types of examination are carried out, both of which are used in current practice:

* Pre-operatively: EOS radiography
* Post-operatively: EOS radiograph and CT scan

Inclusion (m-3; m-1) :

* Patient information at pre-operative visit
* Non-opposition of patient, family member or legal guardian, if applicable
* Questionnaires and clinical examination (standard management)
* EOS during anesthetic consultation

Follow-up visit (m+3):

- Post-operative follow-up consultation EOS and CT scan (1 week prior to visit) + questionnaire and clinical examination

Follow-up visit (m+12):

- Post-operative check-up, questionnaire and clinical examination

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age ≥ 18 years
* Planned surgery: total hip arthroplasty, Minihip or RSA
* Absence of osteoarthritis or osteoarthritis ≤ stage 1 (Tönnis classification) of contralateral hip (Radiographic analysis)
* Patient having given his/her non-opposition to participate in the study
* Patient with social insurance
* Patient willing to comply with all study procedures and duration

Exclusion Criteria:

* Patient with comorbidity(ies) likely to affect biomechanical parameter measurements or surgical conditions:
* Anomalies or anatomical changes of the hip, pelvis or lumbar spine (history of fracture, protrusion, scoliosis, history of orthopedic surgery, dysplasia, torsion disorder)
* Established genetic disease affecting the musculoskeletal system
* Severe or morbid obesity
* Neuromuscular pathologies affecting the limb girdles
* Severe osteoporosis
* Bone location of primary or metastatic cancer (spine, pelvis or femur) - Inequality of lower limb length > 2 cm.
* Minors
* Protected adults
* Pregnant or breast-feeding women
* Administrative reasons: inability to receive informed information, inability to participate in the entire study, lack of social security coverage, refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, primary care clinic at Lille University Hospital, single-center study
Sampling Method: Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Comparing the restoration of femoral hip offset between hip resurfacing procedures (HRP), THA and Minihip-type neck-preserving total hip arthroplasty. | It will be measured using CT scans at 3 months post-op for each hip.
  The primary endpoint will be the difference between the native femoral offset, measured on the healthy contralateral hip, and the postoperative femoral offset of the operated hip. The offset is the distance in millimeters between the axis of the femoral shaft and the center of the femoral head.

SECONDARY OUTCOMES:
Compare the anatomical restoration of frontal and axial parameters between the 3 types of intervention (PTH, Minihip and RSA). | 3 months post-op
  Difference between the contralateral healthy hip and the operated hip at 3 months post-op of the following parameters:
  * frontal parameters: CCD angle (in degrees), limb length, LLL discrepancy (vertical femoral offset in mm), femoral or prosthetic head diameter, acetabulum inclination on the healthy side and cup inclination on the operated side, head-neck ratio (ratio between the diameter of the neck and the head of the femur).
  * axial parameters: femoral or prosthetic neck version, acetabulum version on healthy side and cup version on operated side, total version (neck + acetabulum or cup).
Compare clinical outcomes and patient satisfaction between the 3 procedures (PTH, Minihip and RSA). | 3 months then 1 year post-op
  Variations between the pre-operative and post-operative 3-month and 1-year periods in the following clinical parameters:
  Oxford, Harris, PMA, Devane, UCLA, Forgotten Joint Score Hip (FJS hip), joint amplitudes, ILMI clinical estimate (in cm)
  - Patient satisfaction: measured using a 4-item MCQ (dissatisfied, not very satisfied, satisfied, very satisfied) at 3 months (early recovery) and 1 year (definitive recovery).
Correlate restoration of hip femoral offset and patient functional outcome at 3 months. | 3 months post-op
  Offset restoration, defined as the difference between the native femoral offset, measured on the healthy contralateral hip, and the postoperative femoral offset of the operated hip.
  - Patient functional outcome, defined by the Oxford score.